CLINICAL TRIAL: NCT01944358
Title: Comparisons of Treatment Response to Standard Treatment With Penicillin Between HIV-infected and HIV-uninfected Patients With Syphilis
Brief Title: Comparisons of Serologic Response of Early Syphilis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other); Taichung Veterans General Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); E-DA Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Taiwan HIV and Syphilis study group, National Taiwan University Hospital
Other Study IDs: NTUH rec 201003111R
Record Dates: First submitted 2013-09-07; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Serologic Response of Syphilis; Early Syphilis; High Risk Behavior
Keywords: Syphilis; human immunodeficiency virus; penicillin
MeSH Terms: conditions — Syphilis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Taiwan AIDS study group

SUMMARY:
Syphilis and HIV are prone to occur concomitantly and the two diseases share several modes of acquisition and risk factors such as men who have sex with men (MSM), sexual workers, intravenous drug users, previous history of sexual transmitted diseases (STDs), and multiple partners. HIV infection rates of up to 50% have been reported among patients diagnosed with syphilis in several regions, with higher HIV infection rates among MSM. Besides, syphilis ulcers are proposed to enhance the transmission of HIV. In Taiwan, there is also an increasing prevalence of syphilis and HIV co-infection among MSM. Therefore, to treat syphilis is an important issue for public health.

According to literature review, whether patients with HIV and syphilis co-infection had higher serologic failure rate remains controversial, especially in the era after highly active anti-retroviral therapy (HAART) was introduced since 1996. Ghanem et al recently demonstrated that the use of HAART may reduce syphilis failure rates among HIV-infected patients who have syphilis. In addition, the treatment guideline in 2006 suggested that the treatment of primary syphilis and secondary syphilis is single dose benzathine penicillin G regardless of HIV status; however, it goes on to suggest that "some specialists recommended additional treatments for HIV-infected patients", namely 3 doses, each a week apart. There is no reference and evidence of strength of the suggestion but only specialists' opinion.

In the study, we aim to compare serologic response of syphilis to penicillin treatment between HIV-infected and HIV-uninfected patients and to compare serologic response of early syphilis (primary or secondary) to 1 dose and 3 doses of benzathine penicillin G among HIV-infected patients. A longitudinal follow-up of serologic response will be conducted after syphilis treatment.

ELIGIBILITY:
Inclusion Criteria:

* persons aged ≧20 year-old, who had documented syphilis infection (RPR titer≧ 1:4 and TPPA ≧1:320)

Exclusion Criteria:

* Nil

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persons aged ≧20 year-old, who had documented syphilis infection (RPR titer≧ 1:4 and TPPA ≧1:320)
Sampling Method: Non-Probability Sample
Enrollment: 1128 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To compare serologic response of HIV-infected patients co-infected with early syphilis who received 1-dose or 3-doses benzathine penicillin G | Serial analysis every 6 months. From date of enrollment until the date of first documented treatment failure during 12-months follow up or till the complete of 12-month follow. Final accessed till June, 2013.

SECONDARY OUTCOMES:
To compare the serologic response among HIV-infected and uninfected patients after receiving benzathine penicillin G | Serial analysis every 6 months. From date of enrollment until the date of first documented treatment failure during 12-months follow up or till the complete of 12-month follow. Final accessed till June, 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jui Yang, MD, Principal Investigator — Far Eastern Memorial Hospital; Chien-Chin Hung, PHD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan
  - Far Eastern Memorial Hospital, Taipei, Taiwan